CLINICAL TRIAL: NCT05532137
Title: Effectiveness of a Personalized Intervention Program for the Promotion of the Mediterranean Diet, Based on a Mobile Phone Application (e12HR), in Students of the University of Seville
Brief Title: Effectiveness of an App for Mobile Phones (e-12HR) to Increase Adherence to Mediterranean Diet in University Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Luis María Béjar Prado (Other)
Responsible Party: Sponsor-Investigator, Luis María Béjar Prado, Lecturer (Department of Preventive Medicine and Public Health), University of Seville
Organization: University of Seville (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2813-N-21
Record Dates: First submitted 2022-09-02; First posted 2022-09-08 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Mediterranean Diet; Diet Habits; Healthy Eating Index
Keywords: Mediterranean Diet; Diet Habits; Healthy Eating Index
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Participants (university students) are included by probability single-stage cluster sampling at the Faculties of Medicine and Pharmacy at the University of Seville (Spain), selecting 4 random classrooms in each school.
  Of the 4 selected classrooms in each faculty (Medicine and Pharmacy), 2 are randomly assigned to the control group and 2 to the intervention group.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, participants cannot be blinded. However, the person responsible for the statistical analysis remains blinded throughout the study. In addition, although the different versions of the application are available in the Apple Store or Play Store at all times, personal alphanumeric codes are assigned to the participants; so that each participant only has access to him/her version of the application depending on whether they belong to the intervention group ('feedback' e-12HR) or to the control group ('non-feedback' e-12HR).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): This arm uses the 'non-feedback' e-12HR. This version of the application allows to calculate the Mediterranean Diet Serving Score (MDSS) index.
- Intervention group (Experimental): This arm uses the 'feedback' e-12HR. This version of the application allows to calculate the Mediterranean Diet Serving Score (MDSS) index; additionally, this version is designed to promote the Mediterranean diet.
  Interventions: Behavioral: e-12HR app

INTERVENTIONS:
Behavioral: e-12HR app — The 'feedback' e-12HR version: This version of the application allows to calculate the Mediterranean Diet Serving Score (MDSS) index; additionally, this version is designed to promote the Mediterranean diet with two specific automatic functions:
  1. Evaluation of the user's MDSS index.
  2. Identification of the food groups for which the user has not fulfilled the Mediterranean diet recommendations (in addition, this version also provided the user the consumption recommendations established for these food groups).
  Arms: Intervention group

SUMMARY:
This is a controlled, randomized and multicentric clinical trial aimed at university students and performed at the Faculties of Medicine and Pharmacy at the University of Seville (Spain). Its objective is to evaluate the effect of an intervention based on the use of an information and communication technology (ICT) tool, specifically an application for mobile telephones (called e-12HR), in the improvement of adherence to the Mediterranean diet.

DETAILED DESCRIPTION:
Objective:

To evaluate the effect of an intervention based on the use of an information and communication technology (ICT) tool, specifically an application for mobile telephones (called e-12HR), in the increased adherence to the Mediterranean diet in a population of university students.

Design and setting:

A controlled, randomized and multicentric clinical trial with two parallel groups (control group and intervention group).

Study population:

322 university students (161 participants in each group) are necessary; of both genders, over the age of 18 years, who meet selection criteria.

Study setting:

Faculties of Medicine and Pharmacy at the University of Seville (Spain).

Statistical Analysis Discrete variables are presented as a number followed by percentages. Continuous variables are presented using means and standard deviations.

The data are tested for normality using the nonparametric Kolmogorov-Smirnov test.

Students t-test or the nonparametric Mann-Whitney U-test is used for the analysis of quantitative variables, and the chi-square test is used for the comparison of proportions.

The results are considered significant if p-value < 0.05. Statistical analyses are performed using the SPSS statistical software package ver-sion 26.0 (SPSS Inc., Chicago, Illinois, USA).

Measurements and intervention:

Adherence to the Mediterranean diet is evaluated at seven (baseline), fourteen, twenty-one and twenty-eight days follow-up: the adherence to the Mediterranean diet index selected for the study is the Mediterranean Diet Serving Score (MDSS) index.

The advice on healthy diet recommendations (Mediterranean diet) is common to both groups.

There are two versions of e-12HR in the study: 'feedback' e-12HR and 'non-feedback' e-12HR (both versions of the application allow the collection of data on dietary intake in order to calculate the MDSS index).

Control group: use of 'non-feedback' e-12HR (in order to calculate the MDSS index).

Intervention group: use of 'feedback' e-12HR (in order to calculate the MDSS index; additionally, this version is designed to promote the Mediterranean diet).

ELIGIBILITY:
Inclusion Criteria:

* Both genders.
* Over the age of 18.
* Be a student at the Faculties of Medicine or Pharmacy (University of Seville).
* Possess a mobile telephone with Internet access and iOS or Android operating system.

Exclusion Criteria:

- Chronic pathologies, food intolerances or pregnancy (situations that could require specialized dietary recommendations).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 322 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2024-12-16 (Estimated); Study Completion 2025-12-16 (Estimated)

PRIMARY OUTCOMES:
Change in the total score of the Mediterranean Diet Serving Score (MDSS) index at fourteen days of monitoring in both arms. | To assess the effect of the intervention, the change in the total score of the Mediterranean Diet Serving Score (MDSS) index is calculated at fourteen days after the initial intervention in both arms.
  Mediterranean Diet Serving Score (MDSS) index is a metric which provides an assessment of the degree to which individuals follow the Mediterranean diet. It took into account previously-established rules which consider: Specific food groups, recommendations for consumption frequency for standard servings (per meal, daily or weekly) and a numerical score assigned to each item.
Change in the total score of the Mediterranean Diet Serving Score (MDSS) index at twenty-one days of monitoring in both arms. | To assess the effect of the intervention, the change in the total score of the Mediterranean Diet Serving Score (MDSS) index is calculated at twenty-one days after the initial intervention in both arms.
  Mediterranean Diet Serving Score (MDSS) index is a metric which provides an assessment of the degree to which individuals follow the Mediterranean diet. It took into account previously-established rules which consider: Specific food groups, recommendations for consumption frequency for standard servings (per meal, daily or weekly) and a numerical score assigned to each item.
Change in the total score of the Mediterranean Diet Serving Score (MDSS) index at twenty-eight days of monitoring in both arms. | To assess the effect of the intervention, the change in the total score of the Mediterranean Diet Serving Score (MDSS) index is calculated at twenty-eight days after the initial intervention in both arms.
  Mediterranean Diet Serving Score (MDSS) index is a metric which provides an assessment of the degree to which individuals follow the Mediterranean diet. It took into account previously-established rules which consider: Specific food groups, recommendations for consumption frequency for standard servings (per meal, daily or weekly) and a numerical score assigned to each item.

CONTACTS AND LOCATIONS:
Overall Officials: Luis M Bejar, Doctor, Principal Investigator — Lecturer (Department of Preventive Medicine and Public Health)
Locations (1):
- Department of Preventive Medicine and Public Health, Seville, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bejar LM, Sharp BN, Garcia-Perea MD. The e-EPIDEMIOLOGY Mobile Phone App for Dietary Intake Assessment: Comparison with a Food Frequency Questionnaire. JMIR Res Protoc. 2016 Nov 2;5(4):e208. doi: 10.2196/resprot.5782. PMID 27806922
- [Background] Bejar LM, Vazquez-Limon E. Is there any alternative to traditional food frequency questionnaire for evaluating habitual dietary intake? Nutr Hosp. 2017 Jul 28;34(4):990-888. doi: 10.20960/nh.650. PMID 29095013
- [Background] Bejar LM. First evaluation steps of a new method for dietary intake estimation regarding a list of key food groups in adults and in different sociodemographic and health-related behaviour strata. Public Health Nutr. 2017 Oct;20(15):2660-2669. doi: 10.1017/S1368980017001641. Epub 2017 Aug 9. PMID 28789723
- [Background] Bejar LM, Reyes OA, Garcia-Perea MD. Electronic 12-Hour Dietary Recall (e-12HR): Comparison of a Mobile Phone App for Dietary Intake Assessment With a Food Frequency Questionnaire and Four Dietary Records. JMIR Mhealth Uhealth. 2018 Jun 15;6(6):e10409. doi: 10.2196/10409. PMID 29907555
- [Background] Bejar LM, Garcia-Perea MD, Reyes OA, Vazquez-Limon E. Relative Validity of a Method Based on a Smartphone App (Electronic 12-Hour Dietary Recall) to Estimate Habitual Dietary Intake in Adults. JMIR Mhealth Uhealth. 2019 Apr 11;7(4):e11531. doi: 10.2196/11531. PMID 30973343
- [Background] Bejar LM. Weekend-Weekday Differences in Adherence to the Mediterranean Diet among Spanish University Students. Nutrients. 2022 Jul 8;14(14):2811. doi: 10.3390/nu14142811. PMID 35889767
- [Derived] Bejar LM, Mesa-Rodriguez P, Garcia-Perea MD. Short-Term Effect of a Health Promotion Intervention Based on the Electronic 12-Hour Dietary Recall (e-12HR) Smartphone App on Adherence to the Mediterranean Diet Among Spanish Primary Care Professionals: Randomized Controlled Clinical Trial. JMIR Mhealth Uhealth. 2024 Jan 8;12:e49302. doi: 10.2196/49302. PMID 38190226